CLINICAL TRIAL: NCT02864264
Title: Double-Blind, Randomized, Placebo-Controlled, Single Ascending and Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Target Engagement of BMS-986184 in Healthy Subjects and to Evaluate the Safety, Efficacy, Pharmacokinetics, Target Engagement, and Pharmacodynamics of BMS-986184 in Patients With Moderate to Severe Ulcerative Colitis
Brief Title: Single Ascending Dose and Multiple Ascending Dose Study in Healthy Participants and Proof of Mechanism Study in Patients With Ulcerative Colitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Adverse change in the risk/benefit
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: IM012-004; 2016-000895-72 (EudraCT Number)
Record Dates: First submitted 2016-08-09; First posted 2016-08-11 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Healthy Volunteers; Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Antibodies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Single Ascending Dose (SAD) - IV Panel (Experimental): Single intravenous (IV) dose of BMS-986184 or placebo matching BMS-986184
  Interventions: Drug: BMS-986184; Drug: Placebo matching BMS-986184
- Single Ascending Dose (SAD) - SC Panel (Experimental): Single subcutaneous (SC) dose of BMS-986184 or placebo matching BMS-986184
  Interventions: Drug: BMS-986184; Drug: Placebo matching BMS-986184
- Multiple Ascending Dose (MAD) - IV Panel (Experimental): Multiple IV doses of BMS-986184 or placebo matching BMS-986184
  Interventions: Drug: BMS-986184; Drug: Placebo matching BMS-986184
- Proof of Mechanism (POM) - IV Panel (Experimental): Multiple IV doses of BMS-986184 or placebo matching BMS-986184
  Interventions: Drug: BMS-986184; Drug: Placebo matching BMS-986184

INTERVENTIONS:
Drug: BMS-986184
  Other Names: anti - interferon gamma-induced protein 10(IP-10) antibody
Drug: Placebo matching BMS-986184

SUMMARY:
The primary purpose of this study is to determine if single and multiple doses of BMS-986184 are safe and well tolerated in healthy male and female subjects. The primary purpose of the proof of mechanism study is to determine safety and efficacy in patients with ulcerative colitis.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Women of childbearing potential must have a negative serum pregnancy test within 24 hours prior to the start of study drug
* Diagnosis of ulcerative colitis confirmed by endoscopic and histologic evidence (if no previous confirmation of diagnosis is available or if diagnosis is not conclusive, at time of baseline endoscopy, histology must be performed and read locally to confirm diagnosis)

Exclusion Criteria:

* Any bacterial, fungal or viral infection, including tuberculosis, HIV, hepatitis B or hepatitis C
* Subjects with history of cancer, lymphoproliferative disease, class III or IV congestive heart failure, myocardial infarction, unstable angina pectoris, or any history of significant ocular disease such as glaucoma or retinal disease

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-09-14 (Actual); Primary Completion 2017-09-27 (Actual); Study Completion 2017-09-27 (Actual)

PRIMARY OUTCOMES:
Composite of safety and tolerability of BMS-986184 as assessed by vital sign measurements | Up to 183 days
Composite of safety and tolerability of BMS-986184 as assessed by physical examination findings | Up to 183 days
Composite of safety and tolerability of BMS-986184 as assessed by clinical laboratory test results | Up to 183 days
Composite of safety and tolerability of BMS-986184 as assessed by Electrocardiogram (ECG) assessments | Up to 183 days
Composite of incidence, severity and outcome of all Adverse Events (AEs) | Up to 183 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- Local Institution, Melbourne, Victoria, Australia
- Local Institution, Tbilisi, Georgia
- Local Institution, Chisinau, Moldova

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx